CLINICAL TRIAL: NCT02183428
Title: Relative Bioavailability of BI 1356 and Glyburide After Concomitant Administration of Multiple Oral Doses of BI 1356 5 mg Once Daily and a Single Oral Dose of Glyburide 1.75 mg Compared With the Bioavailability of BI 1356 and Glyburide After Each Treatment Given Alone in Healthy Male and Female Volunteers (an Open Label, Randomised, Two-way Crossover Study of Phase I)
Brief Title: Bioavailability of BI 1356 and Glyburide in Healthy Male and Female Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1218.30
Record Dates: First submitted 2014-07-04; First posted 2014-07-08 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Healthy
MeSH Terms: interventions — Linagliptin; Glyburide

ARMS (2):
- BI 1356 (Experimental): Treatment sequence AB_C or C_AB
  * Treatment A: 5 days of treatment with BI 1356 once per day until steady state followed by
  * Treatment B: 1 day of combined treatment of BI1356 and glyburide
  * Treatment C: 1 day of treatment with glyburide alone
  Interventions: Drug: BI 1356; Drug: Glyburide; Drug: BI 1356 + Glyburide
- Glyburide (Active Comparator): Treatment sequence AB_C or C_AB
  * Treatment A: 5 days of treatment with BI 1356 once per day until steady state followed by
  * Treatment B: 1 day of combined treatment of BI1356 and glyburide
  * Treatment C: 1 day of treatment with glyburide alone
  Interventions: Drug: BI 1356; Drug: Glyburide; Drug: BI 1356 + Glyburide

INTERVENTIONS:
Drug: BI 1356
Drug: Glyburide
Drug: BI 1356 + Glyburide

SUMMARY:
The objective of this study was to investigate the effect of multiple doses BI 1356 given once daily in the estimated highest therapeutic dose of 5 mg until steady state on the pharmacokinetics, safety, and tolerability of a single oral conventional therapeutic dose of 1.75 mg glyburide. In addition, the effect of glyburide as a single oral dose of 1.75 mg being a conventional therapeutic dose on the multiple dose pharmacokinetics of BI 1356 was investigated. Pharmacokinetic profiles of glyburide were determined when given alone or in combination with BI 1356. Pharmacokinetic profiles of BI 1356 and its inactive metabolite CD 1750 were determined at steady state of BI 1356 when given alone or in combination with glyburide.

ELIGIBILITY:
Inclusion Criteria:

* Healthy females and males according to the following criteria: Based upon a complete medical history, including the physical examination, vital signs (Blood Pressure (BP), Pulse Rate (PR)), 12-lead (ECG) Electrocardiogram, clinical laboratory tests
* Age ≥18 and Age ≤55 years
* BMI ≥18.5 and BMI ≤29.9 kg/m2 (Body Mass Index)
* Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice and the local legislation

Exclusion Criteria:

* Any finding of the medical examination (including BP, PR and ECG) deviating from normal and of clinical relevance
* Any evidence of a clinically relevant concomitant disease
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Surgery of the gastrointestinal tract (except appendectomy)
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* History of relevant orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* History of relevant allergy or hypersensitivity (including allergy to drug or its excipients)
* Intake of drugs with a long half-life (> 24 hours) within at least one month or less than 10 half-lives of the respective drug prior to administration or during the trial
* Use of drugs which might reasonably influence the results of the trial or that prolong the QT/QTc interval based on the knowledge at the time of protocol preparation within 10 days prior to administration or during the trial, including herbal products
* Participation in another trial with an investigational drug within two months prior to administration or during the trial
* Smoker (> 10 cigarettes or > 3 cigars or > 3 pipes/day)
* Inability to refrain from smoking on trial days
* Alcohol abuse (more than 60 g/day)
* Drug abuse
* Blood donation (more than 100 mL within four weeks prior to administration or during the trial)
* Excessive physical activities (within one week prior to administration or during the trial)
* Any laboratory value outside the reference range that is of clinical relevance
* Inability to comply with dietary regimen of trial site
* A marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc interval >450 ms)
* A history of additional risk factors for torsade de pointes (e.g., heart failure, hypokalaemia, family history of Long QT Syndrome)
* Galactose intolerance
* Lactase deficiency
* Glucose-galactose-malabsorption

For all female subjects:

* Pregnancy or planning to become pregnant within 2 months of study completion
* Positive pregnancy test
* No adequate contraception e.g. , sterilisation, IUD (intrauterine device), have not been using a barrier method of contraception for at least 3 months prior to participation in the study
* Not willing or unable to use a reliable method of barrier contraception (such as diaphragm with spermicidal cream/jelly or condoms with spermicidal foam), during and up to 2 months after completion/termination of the trial
* Partner is unwilling to use condoms
* Lactation period

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2008-05; Primary Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
AUC0-infinity (area under the concentration-time curve of glyburide in plasma) for several time points | up to 48 hours after drug administration
Cmax (maximum measured concentration of glyburide in plasma) for several time points | up to 48 hours after drug administration
AUCτ,ss (area under the concentration-time curve of the analyte in plasma at steady state over a uniform dosing interval τ) of BI 1356 | up to 48 h after drug administration
Cmax,ss (maximum measured concentration of the analyte in plasma at steady state over a uniform dosing interval τ) of BI 1356 | up to 48 h after drug administration

SECONDARY OUTCOMES:
tmax (time from dosing to the maximum concentration of the analyte in plasma) for several time points | up to 48 hours after drug administration
λz (terminal rate constant in plasma) | up to 48 hours after drug administration
t1/2 (terminal half-life of the analyte in plasma) | up to 48 hours after drug administration
MRTpo (mean residence time of the analyte in the body after po administration) for several time points | up to 48 hours after drug administration
CL/F (apparent clearance of the analyte in the plasma after extravascular administration) for several time points | up to 48 hours after drug administration
Vz/F (apparent volume of distribution during the terminal phase λz following an extravascular dose) for several time points | up to 48 hours after drug administration
Number of patients with adverse events | up to 11 weeks
Assessment of tolerability by investigator on a 4-point scale | Day 1 of treatment B, day 3 of treatment B and C
AUC (area under the concentration-time curve of the analyte in plasma) for several time points | up to 48 h after drug administration
Cmax,ss (maximum measured concentration of the analyte in plasma at steady state over a uniform dosing interval τ) of CD 1750 | up to 48 h after drug administration